CLINICAL TRIAL: NCT04500821
Title: Evaluation of the LipiFlow System With a New Activator (Model LFD-2100)
Brief Title: Evaluation of the LipiFlow System With a New Activator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRYE-105-ACTS
Record Dates: First submitted 2020-07-22; First posted 2020-08-05 (Actual); Results first posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Activator LFD-2100 (Experimental): LipiFlow treatment with the Activators LFD-2100 will be performed on both eyes with MGD
  Interventions: Device: Activator LFD-2100

INTERVENTIONS:
Device: Activator LFD-2100 — LipiFlow treatment with the Activators LFD-2100 will be performed on both eyes with MGD

SUMMARY:
Minimum 50 eyes and up to 100 eyes will be treated in this prospective, open-label clinical study. The investigator or designee will perform LipiFlow treatment with the Activators LFD-2100 on both eyes of a subject. The data from the treatment reports generated by the LipiFlow console and from the questionnaire will be used to assess the clinical utilization of the Activator LFD-2100. This study will be conducted in up to four sites in the USA.

ELIGIBILITY:
Inclusion Criteria:

To be able to participate in this study, subjects must:

* Be at least 22 years old.
* Has been diagnosed as bilateral MGD prior to the study visit, or has evidence of MGD in both eyes. NOTE: MGD diagnosis can be based on prior medical records, investigator opinion or based on assessment of meibomian glands of the lower eyelid.
* Availability, willingness, ability and sufficient cognitive awareness to comply with study protocol, examination procedures and visit.
* Be willing to provide informed consent and authorization to disclose protected health information or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical procedures.
* Ability to understand and respond in English.

Exclusion Criteria:

Subject will not be able to be in the study, if the subject:

* Has a history of certain medical conditions that have been identified as contraindications and precautions of the LipiFlow System
* Has a history of prior eye surgery or trauma, active eye disease, or other eye abnormality in the study eye(s), which in the opinion of the investigator would confound the study results.
* Is pregnant, or is breast feeding.
* Concurrent participation or expected participation in an interventional (i.e., surgical or pharmaceutical interventional) clinical trial within 14 days prior to study screening.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision Clinical Trials, Study Director — Johnson & Johnson Surgical vision
Locations (3):
- United States (3):
  - Empire Eye and Laser Center, Bakersfield, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Texas Eye Research Center, Hurst, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 88 eyes of 44 subjects with meibomian gland dysfunction were enrolled.
Units Other Than Participants: Eyes
Groups:
- Activator LFD-2100: Lipiflow treatment with Activator LFD-2100
Period: Overall Study
Arm/Group | Activator LFD-2100
Started | 44; 88 Eyes
Completed | 44; 88 Eyes
Not Completed | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Arm/Group | Activator LFD-2100
Number analyzed (Participants) | 44
Age, Customized [Number; unit: Participants]
  < 30 years | 0
  30-39 years | 0
  40-49 years | 1
  50-59 years | 6
  60-69 years | 19
  >= 70 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 31
  Sex: Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 3
  Ethnicity: Not Hispanic or Latino | 41
  Ethnicity: Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 2
  Black | 0
  Native Hawaiian/Pacific Islander | 0
  Caucasian | 42

OUTCOME MEASURES:

1. Primary Outcome: Successful Completion of LipiFlow Treatment With Activator LFD-2100
Description: Evaluation of the clinical use of the LipiFlow system with the Activator LFD-2100
Time Frame: 1 day after completion of LipiFlow treatment
Population: All treated eyes
Measure: Number (95% Confidence Interval); unit: Percent of eyes
Units Other Than Participants: Eyes
Arm/Group | Activator LFD-2100
Number analyzed (Participants) | 44
Number analyzed (Eyes) | 88
Percent of eyes | 100 [96 to 100]

ADVERSE EVENTS:
Time Frame: During the course of the study until completion, 1 up to 2 days.
Description: Analysis population include all eyes (88 eyes) of 44 participants treated with Lipiflow with Activator LFD-2100. All adverse events (AEs), ocular and non-ocular, were monitored/assessed and planned to be reported for each eye separately.
Groups:
- Right Eye (OD); Left Eye (OS): LipiFlow treatment with Activator LFD-2100
Arm/Group | Right Eye (OD) | Left Eye (OS)
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review results communication prior to public release and can embargo communications regarding trial results at anytime.

DOCUMENTS (2):
  • Study Protocol (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/21/NCT04500821/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT04500821/SAP_001.pdf